CLINICAL TRIAL: NCT06874907
Title: First Trimester Prediction of Gestational Diabetes Mellitus by Continuous Glucose Monitoring.
Acronym: GLUCO-GCM
Status: Recruiting | Type: Observational
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IMIB-GLC-2023-03
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Continuous glucose monitoring: First trimester prediction of gestational diabetes mellitus by continuous glucose monitoring
  Interventions: Procedure: Glucose monitoring

INTERVENTIONS:
Procedure: Glucose monitoring — Glucose monitoring

SUMMARY:
Gestational diabetes mellitus (GDM) is the most common complication of pregnancy, with an incidence rate of 10-15% [1]. Common risk factors for GDM are increased maternal age and weight and as a consequence of women delaying childbirth and increasing incidence of obesity, there is a corresponding increase in the rate of GDM. GDM is associated with an increased risk of maternal and perinatal short and long-term complications . These include macrosomia, shoulder dystocia, neonatal hypoglycaemia, neonatal hyperbilirubinemia, and perinatal mortality. Maternal complications include higher risks of hypertensive disorders, perineal trauma, and caesarean section. Additionally, both the mothers with GDM and their infants have an increased risk of developing type 2 diabetes mellitus and cardiovascular disease later in life .

Screening and diagnosis of GDM is currently based on an oral glucose tolerance (OGTT), which is carried out at 26-28 weeks' gestation. In addition, an OGTT is carried out at 11-13 weeks in women considered to be at increased risk of GDM based on their demographic characteristics and medical history. Screening and diagnosis of GDM is traditionally delayed until the late second or early third trimester of pregnancy with the rationale that the diabetogenic effects of pregnancy increase with gestation and therefore delayed testing would maximize the detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18 years
* Planned antenatal care at the same centre (i.e. not planning to move before delivery).
* Singleton pregnancy.
* Informed and written consent.

Exclusion Criteria:

* Age <18 years;
* Multiple pregnancy in current pregnancy;

  * Unconscious or very ill; · Serious mental illness;
  * Learning difficulties;
  * Not fluent in local language and absence of interpreter;
  * Severe congenital anomaly on ultrasound;
  * Pre-existing diabetes mellitus type 1 or 2;
  * Patients undergoing metformin therapy for infertility.
  * Significant pre-pregnancy comorbidities that increase risk in pregnancy, for example renal failure, severe liver disease, transplantation, cardiac failure, psychiatric conditions requiring in-patient admission (<1 year);
  * Significant co-morbidity in the current pregnancy, nephropathy (estimated GFR <60ml/min), other physical or psychological conditions likely to interfere with the conduct of the study and/or interpretation of the trial results;
  * Participating in another intervention study that influences outcomes of this study;
  * Allergy to adhesive materials;
  * Allergy to any of the components of the glucose test:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy women
Study Population: Pregnant patients over 18 years of age
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Value of CGM (Continuous glucose monitoring) at 12 and 28 weeks of gestation in the prediction of GDM (Gestational diabetes mellitus ) | Up to 28 weeks
  GDM is defined by abnormal results of 75mg OGTT(Oral Glucose Tolerance Test) at 28 weeks' gestation

SECONDARY OUTCOMES:
Number of patients with Gestational hypertension | Up to 28 weeks
  blood pressure readings are higher than 140/90 mm Hg in a woman who had normal blood pressure prior to 20 weeks and has no proteinuria (excess protein in the urine)
Glycaemic profile according to CGM (Continuous glucose monitoring)at 12 and 28 weeks and OGTT(Gestational diabetes mellitus ) results at 28 weeks | Up to 28 weeks
  Number of patients with Delivery by caesarean section
Glycaemic profile according to CGM (Continuous glucose monitoring)at 12 and 28 weeks and OGTT(Gestational diabetes mellitus ) results at 28 weeks | Up to 28 weeks
  Number of patients with Stillbirth, neonatal death, perinatal death
Glycaemic profile according to CGM (Continuous glucose monitoring)at 12 and 28 weeks and OGTT(Gestational diabetes mellitus ) results at 28 weeks | Up to 28 weeks
  Number of patients with Large for gestational age neonate (>90th and 95th percentile for gestation)
Glycaemic profile according to CGM (Continuous glucose monitoring)at 12 and 28 weeks and OGTT(Gestational diabetes mellitus ) results at 28 weeks | Up to 28 weeks
  Number of patients with Neonatal hyperglycaemia
Glycaemic profile according to CGM (Continuous glucose monitoring)at 12 and 28 weeks and OGTT(Gestational diabetes mellitus ) results at 28 weeks | Up to 28 weeks
  Number of patients with Neonatal hyperbilirubinemia
Glycaemic profile according to CGM (Continuous glucose monitoring)at 12 and 28 weeks and OGTT(Gestational diabetes mellitus ) results at 28 weeks | Up to 28 weeks
  Number of patients with Neonatal unit (NNU) admission for ≥48 hours
Glycaemic profile according to CGM (Continuous glucose monitoring)at 12 and 28 weeks and OGTT(Gestational diabetes mellitus ) results at 28 weeks | Up to 28 weeks
  Number of days (Length of stay) in the Neonatal Intensive Unit.

CONTACTS AND LOCATIONS:
Overall Officials: Catalina de Paco Matallana, MD, Principal Investigator — HCUVA
Locations (1):
- HCUVA, El Palmar, Murcia, Spain